CLINICAL TRIAL: NCT04980105
Title: Intra-articular Injections of Platelet-rich Plasma, Hyaluronic Acid, or Corticosteroids for Knee Osteoarthritis, Which is Better? A Prospective Study of a Single-blind Randomized Control Trial RCT From the Iraqi Population
Brief Title: Intra-articular Injections of Platelet-rich Plasma, Hyaluronic Acid, or Corticosteroids for Knee Osteoarthritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Wasit (Other)
Responsible Party: Principal Investigator, Usama Al-Sari, Senior Lecturer of Rheumatology M.B.,Ch.B, MSc , PhD, University of Wasit
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UOW/MS102
Record Dates: First submitted 2021-07-07; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid; Methylprednisolone Acetate

STUDY DESIGN:
Intervention Model Description: A total of 150 participants fulfilling the inclusion criteria, patients were randomly assigned into three groups by a computer-based protocol. The patients were separated into three groups according to the type of treatment administered.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Platelet-rich plasma arm (Experimental)
  Interventions: Biological: Platelet-rich plasma
- Hyaluronic acid arm (Active Comparator)
  Interventions: Drug: Hyaluronic acid
- Methylprednisolone acetate arm (Active Comparator)
  Interventions: Drug: Methylprednisolone acetate injectable suspension (DEPO-MEDROL®)

INTERVENTIONS:
Biological: Platelet-rich plasma — Two intra-articular injections of autologous platelets-rich plasma (PRP) in two weeks intervals between the first and the second injection.
  Arms: Platelet-rich plasma arm
Drug: Hyaluronic acid — Two intraarticular injections of hyaluronic acid (60 mg) in two weeks intervals between the first and the second injection
  Arms: Hyaluronic acid arm
Drug: Methylprednisolone acetate injectable suspension (DEPO-MEDROL®) — Single methylprednisolone acetate intraarticular injection (DEPO-MEDROL® pfizer 80 mg) mixed with 3cc of (xylocaine 2% concentration)
  Arms: Methylprednisolone acetate arm

SUMMARY:
To assess if there are any differences among platelet-rich plasma, hyaluronic acid, and corticosteroid knee intra-articular injection regarding function and pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 35-65 years old
* Patient with knee pain that had been continuing for at least 12 months with no relief using anti-inﬂammatory medications and that deteriorated with weight-bearing
* Knee osteoarthritis that classified as mild-moderate or moderate-severe (Kellgren-Lawrence Grade 2, 3, or 4)

Exclusion Criteria:

* Age > 65 years
* The recent history of knee trauma
* Autoimmune rheumatic diseases
* Accompanying severe hip OA
* Thrombocytopenia or other blood diseases
* Immunosuppressive or anticoagulant treatment
* The invasive procedure applied to the knee
* Intra-articular steroid injection to the knee within the previous 12 months
* Previous joint infection
* Uncontrolled systemic diseases such as diabetes or hypertension, and cancer
* Excessive varus/valgus knee deformity

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go test (TUG) | 18th months
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turn around 180 degrees, walk back to the chair, and sit down while turning 180 degrees
Visual Analogue Scale (VAS) | 18th months
  The VAS uses a straight 10 centimeter line with one end being 'no pain' and on the other end the 'worst imaginable pain'. The patient chooses a spot on the line then places a perpendicular line to indicate their pain level

CONTACTS AND LOCATIONS:
Overall Officials: Usama A Al-Sari, PhD, Principal Investigator — UOW
Locations (1):
- University of Wasit, Wāsiţ, Iraq